CLINICAL TRIAL: NCT04514588
Title: Associations Between Genetic Markers of Caffeine Metabolism, Appetite Hormones and Body Weight
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Gkouskou Kalliopi (Other)
Responsible Party: Sponsor-Investigator, Gkouskou Kalliopi, Dr Kalliopi Gkouskou principal investigator, National and Kapodistrian University of Athens
Organization: National and Kapodistrian University of Athens (Other)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: AP336.30.06.2020
Record Dates: First submitted 2020-08-02; First posted 2020-08-17 (Actual); Last update posted 2020-08-17 (Actual); Status verified 2020-08

CONDITIONS: Food Consumption and Appetite; Food Habits; Caffeine
MeSH Terms: conditions — Feeding Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- caffeine consumption and metabolism (Other): Participants will take part in two trials. Each trial will last one day at least one week apart. During the first trial half of the participants will consume caffeine (5mgr/kgr) and the rest only water. During the second trial a crossover design will be applied
  Interventions: Dietary Supplement: caffeine consumption
- control (Other): Control group will consume only water (not coffee) and the same parameters will be recorded as previously
  Interventions: Dietary Supplement: caffeine consumption

INTERVENTIONS:
Dietary Supplement: caffeine consumption — In this trial we are going to study the results of the consumption of 5mgr/kgr body weight of caffeine on appetite, food consumption and hormones ghrelin, asprosin, leptin and pancreatic polypeptide in relation to gene polymorphisms that affect caffeine metabolism and body weight

SUMMARY:
The effect of caffeine on appetite and body weight is controversial. Mostly epidemiological studies exist that show either a negative effect (reduction of appetite and body weight) or no effect. In this trial we are going to study the results of the consumption of 5mgr/kgr body weight of caffeine on appetite, food consumption and hormones ghrelin, asprosin, leptin and pancreatic polypeptide in relation to gene polymorphisms that affect caffeine metabolism and body weight. Seventy subjects will participate in a cross sectional study consisting of two trials (with or without the consumption of caffeine) in order to study the aforementioned parameters. Differences of total calories consumption between fast metabolizers of caffeine and the rest of the participants is the primary outcome.

DETAILED DESCRIPTION:
In more detail, participants will be recruited through local advertisements in the university campus so that to be of normal weight (BMI<25) and apparently healthy. Smokers, special population groups, i.e. athletes, pregnant women etc., those having a chronic or acute disease and those on medication will be excluded from the study.

Experimental protocol. Each volunteer will take part in 2 trials (with 7days interval between them) in a random order (using a random-number table). Female participants will be on the follicular phase of their menstrual cycle during the experiments to avoid variability in appetite [doi.org/10.1016/j.appet.2018.01.029.]. The week preceding each experimental day, participants will be instructed to abstain from any caffeine. Furthermore, the day preceding each experimental day participants will be instructed to abstain from alcohol source and physical exercise, to get enough sleep (~7 h) and to come to the lab after an overnight fast of 10 h. Furthermore, the days before the experiment, volunteers will be asked to consume similar foods and quantities, keeping more or less constant eating patterns. Participants will arrive at the lab in the morning 9 am after an overnight fast of 10 h. They will consume a breakfast snack along with one of the three experimental drinks within 5 min. The snack will consist of 1 slice of white bread, 5 g of butter and 10 g of white sugar, providing 142 kcal (6.5% of energy from proteins, 62.5% from carbohydrates and 31.0% from lipids). The experimental drinks will be either (a) 200 mL of instant coffee providing 5 mg caffeine/kg body weight or (b) 200 mL of water (Control). After a 3-h period, participants will be offered an ad libitum lunch meal from a buffet, consisting of common Greek diet foods (pasta, tomato sauce, beef, salad, cheese, yogurt, fruit and juice). They will be instructed to consume as much food as they desire until they feel satiated, within 30 min. Researchers will record the exact amount of food consumed by weighting the foods that will be chosen and their remnants. In addition, a detailed recording of the foods participants are going to consume later in the evening will be performed from a registered dietician through recall questionnaires.

Molecular and biochemical parameters that are going to be recorded with the utilization of standardized generally accepted protocols are blood pressure, body weight and other anthropometric parameters, blood levels of ghrelin, asprosin, leptin, pancreatic polypeptide, insulin and glucose, and genetic markers that are related to caffeine metabolism (CYP1A2 rs2069514 και CYP1A2 rs762251), as well as to an obesity genetic risk score (32SNPs).

Primary and secondary outcomes Based on genotype data, participants will be categorized as fast, medium and slow metabolizers of caffeine. For sample size calculation differences of total calories consumptions between groups will be utilized as primary outcome. More specifically, since a small participation of slow metabolizers are expected, these subjects will be grouped together with medium metabolizers. A difference of total calories consumption that exceeds 20% between the two groups is considered clinically significant. Taking into account an attrition rate of 10% between the two trials (caffeine and control) a total of about 70 participants are required for the study.

Macronutrients (protein, carbohydrates and lipids) consumption, responses on visual analog scales for satiety and appetite, hormones concentrations will be studied as secondary outcomes

ELIGIBILITY:
Inclusion Criteria:

* normal weight (BMI<25)
* apparently healthy participants

Exclusion Criteria:

* smokers,
* special population groups, i.e. athletes, pregnant women etc.,
* people with a chronic or acute disease and
* those on medication

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 70 (Estimated)
Dates: Start 2020-06-30 (Actual); Primary Completion 2022-06-30 (Estimated); Study Completion 2022-06-30 (Estimated)

PRIMARY OUTCOMES:
total calories consumption change | two trials (caffeine and control) two weeks apart each lasting one day
  a detail recording of foods and their quantities during the day of the trial will take place

SECONDARY OUTCOMES:
hormones concentrations change | two trials (caffeine and control) two weeks apart each lasting one day
  insulin, ghrelin, asprosin, leptin and pancreatic polypeptide
VAS (visual analog scale-11-likert scale with greater numbers indicating greater appetite) change for appetite | two trials (caffeine and control) two weeks apart each lasting one day
  visual analog scales administered in specific time frames 15 min before and 15, 30, 60, 90, 120, 150, 180 min after the consumption of breakfast with or without caffeine
VAS (visual analog scale 11-likert scale with greater numbers indicating greater satiety) change for satiety | two trials (caffeine and control) two weeks apart each lasting one day
  visual analog scales administered in specific time frames 15 min before and 15, 30, 60, 90, 120, 150, 180 min after the consumption of breakfast with or without caffeine
various macronutrients consumption change | two trials (caffeine and control) two weeks apart each lasting one day
  a detail recording of foods and their quantities during the day of the trial will take plac

CONTACTS AND LOCATIONS:
Overall Officials: Aristides Eliopoulos, prof, Study Chair — University of Athens
Locations (1):
- University of West Attica, Aigáleo, Attica, Greece

REFERENCES:
- [Derived] Gkouskou KG, Georgiopoulos G, Vlastos I, Lazou E, Chaniotis D, Papaioannou TG, Mantzoros CS, Sanoudou D, Eliopoulos AG. CYP1A2 polymorphisms modify the association of habitual coffee consumption with appetite, macronutrient intake, and body mass index: results from an observational cohort and a cross-over randomized study. Int J Obes (Lond). 2022 Jan;46(1):162-168. doi: 10.1038/s41366-021-00972-6. Epub 2021 Sep 25. PMID 34564706